CLINICAL TRIAL: NCT04425408
Title: Randomized Cross Over Trial Assessing the Efficacy of Two Different Positional Therapies for Positional Obstructive Sleep Apnea (POSA)
Brief Title: Comparison of 2 Different Positional Therapies for Positional Obstructive Sleep Apnea Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to recruit
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Deputy Head of the Respiratory Unit, Clinical Professor, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B076201941938
Record Dates: First submitted 2020-02-05; First posted 2020-06-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Positional Obstructive Sleep Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional pillow followed by vibrating belt (Experimental): 26 patients with positional sleep apnea will be randomized to spend 3 nights using a positional pillow followed by a vibrating belt. The time spend on supine position will be monitored on each device and a satisfaction questionnaire as well as a sleep quality questionnaire will be performed after the use of each device.
  Interventions: Device: Consecutive trial of two different devices for the treatment of positional sleep apnoea, for 3 nights with each device (positional pillow and vibrating belt).
- Vibrating belt followed by positional pillow (Experimental): 26 patients with positional sleep apnea will be randomized to spend 3 nights using a vibrating belt followed by a positional pillow. The time spend on supine position will be monitored on each device and a satisfaction questionnaire as well as a sleep quality questionnaire will be performed after the use of each device.
  Interventions: Device: Consecutive trial of two different devices for the treatment of positional sleep apnoea, for 3 nights with each device (positional pillow and vibrating belt).

INTERVENTIONS:
Device: Consecutive trial of two different devices for the treatment of positional sleep apnoea, for 3 nights with each device (positional pillow and vibrating belt). — Patients will be randomly allocated to use either a positional pillow or a vibrating belt for three consecutive nights at home followed by three nights with the other device.

SUMMARY:
The proposed study is a randomized cross over trial assessing the efficacy of two different positional therapies for positional obstructive sleep apnea (POSA).

The effectiveness of the two different therapeutic devices (Positional pillow and vibrating belt) in reducing the time spent sleeping supine, and therefore at risk of apnoeas, will be evaluated consecutively in 52 subjects with a de novo diagnosis of positional sleep apnoea.

The subjective quality of sleep will also be evaluated prior to treatment and following the use of each separate device by means of a "Quality of sleep questionnaire"

DETAILED DESCRIPTION:
Patients with a de novo diagnosis of positional sleep apnoea on a polysomnography performed in our sleep lab will be asked to participate to the study. They should fulfill the Mador definiton of POSA.

A home recording of sleep position with Somnibel Pro will be conduted for 2 consecutive nights. In case of confirmation of supine sleep at home (Mean supine sleep >30% of total sleep time) the patient will be asked to use two different positional therapy devices consecutively (Positional pillow and vibrating belt), 3 nights each, in a random order, with concomitant recording of sleep position with the Somnibel Pro. Global satisfaction questionnaire will be assessed by a simple visual analogic scale (is it easy to use? Is it confortable? Is it efficient on snoring? Is it efficient on sleep apnea? Would you pay for such treatment? Willingness to use it on a long-term basis?) The subjective sleep quality will also be assessed by means of "Sleep quality questionnaire", prior to commencing treatment, and consecutively after 3 nights on each individual therapy.

Statistical analysis:

Efficacy of Positional pillow (Posiform) and vibrating belt (Somnofit) Percentage sleep on back on treatment will be compared to mean percentage sleep on back without treatment, at home, for both devices. Comparison on surrogate AHI based on diagnostic polysomnography, with and without each device. Global satisfaction with the devices will also be compared between devices.

The sleep quality will be compared on the two devices using the "Sleep quality questionnaire".

The sample size of 52 subjects (26 in each arm), has been calculated to obtain a power of 90% and allow a drop out rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients able to give writtent consent with a de novo diagnosis of positional sleep apnoea according to a polysomnograph.

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of supine sleep time without treatment and between the two devices (positional pillow and vibrating belt). | 5 years
  The percentage of supine sleep on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- Centre hospitalier universitaire Saint Pierre, Rue Haute 322, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No